CLINICAL TRIAL: NCT03211507
Title: Idiopathic Pulmonary Fibrosis Job Exposures Study
Acronym: IPFJES
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Wellcome Trust (Other); University Hospital Southampton NHS Foundation Trust (Other); Imperial College Healthcare NHS Trust (Other); Heart of England NHS Foundation Trust (Unknown); Liverpool University Hospitals NHS Foundation Trust (Other Government); Papworth Hospital NHS Foundation Trust (Other Government); Nottingham University Hospitals NHS Trust (Other); University Hospital of South Manchester (Unknown); Guy's and St Thomas' NHS Foundation Trust (Other); North Bristol NHS Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Royal Devon and Exeter NHS Foundation Trust (Other); Somerset NHS Foundation Trust (Other); Royal Infirmary of Edinburgh (Other); Morriston Hospital (Unknown); Aberdeen Royal Infirmary (Other); Worcestershire Acute Hospitals NHS Trust (Other); University Hospital Birmingham NHS Foundation Trust (Other); Portsmouth Hospitals NHS Trust (Other Government); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); Glasgow Royal Infirmary (Other)
Responsible Party: Sponsor
Other Study IDs: 16SM3627
Record Dates: First submitted 2017-05-02; First posted 2017-07-07 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: IPF; Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Males with an incident diagnosis of IPF made between the 1st of February 2017 and the 5th of October 2019.
  Interventions: Other: Computer-assisted telephone interview; Genetic: Genetic analysis
- Controls: Males with an incident hospital outpatient attendance between the 1st of February 2017 and the 5th of October 2019 who do not have a diagnosis of IPF. At each participating centre a control clinic is randomly selected from all control clinics that the research team is able to recruit from; this clinic is the source clinic for controls for the duration of the study.
  Interventions: Other: Computer-assisted telephone interview; Genetic: Genetic analysis

INTERVENTIONS:
Other: Computer-assisted telephone interview — Occupational history
Genetic: Genetic analysis — To include analysis of known susceptibility markers

SUMMARY:
A case-control study to investigate whether job exposures are an under-recognized cause of idiopathic pulmonary fibrosis (IPF) using an interview to collect information about previous jobs and a blood test to investigate genetic susceptibility.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a scarring lung disease. It damages the air sacs that allow oxygen to be transferred into the blood and transported to vital organs. These changes make people with IPF cough and feel short of breath. It not known what causes the damage. People who get IPF are usually older than 40; it's a very serious illness that cannot be cured and gets worse over time. Statistics show that IPF is becoming more common in the UK but it's not known why. It can be difficult for doctors to tell if someone has IPF or another disease called asbestosis.

ELIGIBILITY:
For cases

Inclusion Criteria:

* New diagnosis of IPF between February 2017 and October 2019

Exclusion Criteria:

* Unable to give informed consent
* Ever worked outside of the UK

For controls

Inclusion Criteria:

* New outpatient department attendee between February 2017 and October 2019

Exclusion Criteria:

* Unable to give informed consent
* Ever worked outside of the UK (does not include work outside the UK by members of the armed forces or merchant navy)
* Diagnosis of IPF

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital based
Sampling Method: Probability Sample
Enrollment: 960 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2019-10-05 (Actual)

PRIMARY OUTCOMES:
Association between asbestos exposure and IPF | 2 years
  estimated using logistic regression for any vs no asbestos exposure and adjusting for age and smoking status

SECONDARY OUTCOMES:
Dose-response relationship between asbestos exposure and IPF | 2 years
  estimated using logistic regression for categories of cumulative exposure and adjusting for age and smoking status
Gene-environment interaction (for MUC5B rs35705950 and asbestos exposure) odds ratio. | 2 years
  MUC5B rs35705950 and asbestos exposure odds ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Reynolds, Study Director — Imperial College London
Locations (1):
- Imperial Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reynolds CJ, Sisodia R, Barber C, Moffatt M, Minelli C, De Matteis S, Cherrie JW, Newman Taylor A, Cullinan P. What role for asbestos in idiopathic pulmonary fibrosis? Findings from the IPF job exposures case-control study. Occup Environ Med. 2023 Feb;80(2):97-103. doi: 10.1136/oemed-2022-108404. Epub 2023 Jan 12. PMID 36635100
- See also: Full study documentation — https://github.com/drcjar/ipfjes/blob/master/README.md